CLINICAL TRIAL: NCT01148836
Title: Coenzyme Q-10 in the Treatment of Pulmonary Arterial Hypertension
Brief Title: Coenzyme Q-10 and Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Jacqueline Sharp, Nurse Practitioner, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-497
Record Dates: First submitted 2010-03-19; First posted 2010-06-22 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Coenzyme Q-10; Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension Class I (Venice 2003)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Ubiquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coenzyme Q 10 and Pulmonary Hypertension (Experimental): PAH subjects to take Co-Q daily for three months
  Interventions: Dietary Supplement: Coenzyme Q-10 in Pulmonary Hypertension subjects
- Coenzyme Q 10 and Normal Controls (Experimental): Normal controls to take Co-Q daily for three months
  Interventions: Dietary Supplement: Coenzyme Q-10 in Normal Control subjects

INTERVENTIONS:
Dietary Supplement: Coenzyme Q-10 in Pulmonary Hypertension subjects — Take 100mg Co-Q for three times daily
  Other Names: Coenzyme Q: Nutritional Supplement
  Arms: Coenzyme Q 10 and Pulmonary Hypertension
Dietary Supplement: Coenzyme Q-10 in Normal Control subjects — Take 100mg Co-Q for three times daily
  Arms: Coenzyme Q 10 and Normal Controls

SUMMARY:
The purpose of this study is to evaluate the effects of Coenzyme Q-10, an antioxidant, in the treatment of pulmonary hypertension.

DETAILED DESCRIPTION:
Abnormalities in the blood vessels in the lung are the hallmark of pulmonary hypertension. Links between increased free radical production, mitochondrial dysfunction and pulmonary hypertension have been studied but are poorly understood. The mitochondria of cells is the location where cellular energy is created and free radicals are atoms or groups of atoms with an odd (unpaired) number of electrons and can be formed when oxygen interacts with certain molecules. Once formed these reactive radicals can start a chain reaction, like dominoes. Their chief danger comes from the damage they can do when they react with important cellular components. Cells may function poorly or die if this occurs. The body produces free radicals in the normal course of energy production and in pulmonary hypertension, free radical production is found to be increased. To prevent free radical damage the body has a defense system of antioxidants. Coenzyme Q-10 is an antioxidant and it helps to protect cells from damage caused by the body's own free radicals. By providing oral supplementation of coenzyme Q-10, free radical levels will be decreased and cellular functioning in the pulmonary blood vessels may improve and even return to near normal functioning.

The purpose of this study is to evaluate the effects of coenzyme Q-10, an antioxidant, in the treatment of pulmonary hypertension. We will assess coenzyme Q-10 supplementation in the treatment of pulmonary hypertension by clinical measurements and blood levels of certain cellular components. We would like to assess the effects of coenzyme Q-10 on the pulmonary vessels by measuring the lung diffusing capacity (a breathing test) and exhaled Nitric Oxide (NO) (a substance in the body that relaxes or dilates blood vessels). We will also measure endothelial progenitor cells (cells from the bone marrow) from a blood sample; these cells are markers of measure of blood vessel formation and repair. We will also measure the activity of superoxide dismutase (a protein in cells that executes the breakdown of a free radical into oxygen and hydrogen peroxide) in the blood. In addition, we will measure levels of coenzyme Q-10 in the blood. Other markers of disease response to therapy will be done including physical exam, BNP level (a blood marker that correlates with heart function), 6-minute walk and echocardiography (ultrasound of the heart). A total of 60ml (5 tablespoons) of blood will be drawn at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age equal to or greater than 18 not to exceed 65.
* Patients with PAH Class 1 (Venice 2003)
* PAH medications must not have changed for the last two months.
* Women of child-bearing age must use a double-barrier local contraception until completion of study.
* Subjects must demonstrate understanding of study and sign informed consent and have a reliable method of communication for contact and the ability to comply with the study requirements.

Exclusion Criteria:

* Participation in any other studies at the time of enrollment
* History of any significant illness within four weeks of starting Coenzyme Q-10
* Hepatic insufficiency (transaminase levels >4 fold the upper limit of normal or bilirubin >2 fold the upper limit of normal).
* Renal insufficiency (creatinine >2)
* Pregnancy,breast-feeding or lack of safe contraception.
* Acute heart failure
* Known allergy to the study drug or drugs similar to the study drug
* History of drug or alcohol abuse within last 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Sharp, CNP, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | Pulmonary Hypertension Subjects (Disease)
Started | 8 (Enrollment completed) | 10
Completed | 7 (Enrollment completed) | 8
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls Subjects | Pulmonary Hypertension Subjects | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (5) | 41 (3) | 41.5 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular End Diastolic Volume
Description: Amount of blood in ventricle at end of diastole
Time Frame: before and after three months of CoQ
Population: Due to financial constraints only PAH subjects had echocardiograms performed before and after Co-Q
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Pulmonary Hypertension Subjects: Pulmonary Hypertension subjects taking Co-Q for three months
Arm/Group | Pulmonary Hypertension Subjects
Number analyzed (Participants) | 8
ml
  Before Co-Q | 81 (10)
  After Co-Q | 70 (8)

2. Primary Outcome: Right Ventricular Outflow
Description: Velocity time interval
Time Frame: before and after three months of CoQ
Population: Due to financial constraints only PAH subjects had echocardiograms performed before and after Co-Q
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pulmonary Hypertension Subjects
Number analyzed (Participants) | 8
cm
  Before Co-Q | 11.3 (1.4)
  After Co-Q | 13.5 (1.6)

3. Primary Outcome: Right Ventricle Myocardial Performance
Description: Tei Index=(IRT+ICT)/ET, where IRT is isovolumic
Time Frame: before and after three months of CoQ
Population: Due to financial constraints only PAH subjects had echocardiograms performed before and after Co-Q
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pulmonary Hypertension Subjects
Number analyzed (Participants) | 8
ratio
  Before Co-Q | 0.9 (0.2)
  After Co-Q | 0.7 (0.1)

4. Primary Outcome: Tricuspid Regurgitation Grade
Description: Tricuspid Regurgitation Grade ranges from 1 (normal) to 4 (severe regurgitation)
Time Frame: before and after three months of CoQ
Population: Due to financial constraints only PAH subjects had echocardiograms performed before and after Co-Q
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulmonary Hypertension Subjects
Number analyzed (Participants) | 8
units on a scale
  Before Co-Q | 1.4 (0.3)
  After Co-Q | 1.2 (0.3)

5. Primary Outcome: Right Atrial Pressure
Time Frame: before and after three months of CoQ
Population: Due to financial constraints only PAH subjects had echocardiograms performed before and after Co-Q
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pulmonary Hypertension Subjects
Number analyzed (Participants) | 8
mmHg
  Before Co-Q | 10 (2)
  After Co-Q | 8 (1)

6. Secondary Outcome: Red Blood Cells
Time Frame: before and after three months of CoQ
Measure: Mean (Standard Deviation); unit: 10^6 cells/µl
Groups:
- Normal Controls: Normal controls taking Co-Q for three months
Arm/Group | Pulmonary Hypertension Subjects | Normal Controls
Number analyzed (Participants) | 8 | 7
10^6 cells/µl
  Before Co-Q | 5.2 (0.2) | 4.5 (0.1)
  After Co-Q | 5.2 (0.2) | 4.3 (0.2)

7. Secondary Outcome: Hemoglobin
Time Frame: before and after three months of CoQ
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Pulmonary Hypertension Subjects | Normal Controls
Number analyzed (Participants) | 8 | 7
g/dl
  Before Co-Q | 14.1 (0.9) | 13.3 (0.4)
  After Co-Q | 14.6 (0.8) | 12.9 (0.5)

8. Secondary Outcome: Hematocrit
Time Frame: before and after three months of CoQ
Measure: Mean (Standard Deviation); unit: % of red blood cell
Arm/Group | Pulmonary Hypertension Subjects | Normal Controls
Number analyzed (Participants) | 8 | 7
% of red blood cell
  Before Co-Q | 43.0 (2.1) | 39.9 (1.0)
  After Co-Q | 43.8 (1.8) | 38.6 (1.3)

9. Secondary Outcome: Mean Corpuscular Hemoglobin
Time Frame: before and after three months of CoQ
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Pulmonary Hypertension Subjects | Normal Controls
Number analyzed (Participants) | 8 | 7
pg
  Before Co-Q | 26.8 (1.1) | 29.9 (0.8)
  After Co-Q | 27.8 (1.0) | 29.9 (0.7)

10. Secondary Outcome: Red Blood Cell Distribution Width
Time Frame: before and after three months of CoQ
Measure: Mean (Standard Deviation); unit: percentage of sizes of red blood cells
Arm/Group | Pulmonary Hypertension Subjects | Normal Controls
Number analyzed (Participants) | 8 | 7
percentage of sizes of red blood cells
  Before Co-Q | 15.0 (0.6) | 12.9 (0.2)
  After Co-Q | 14.5 (0.5) | 12.9 (0.4)

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over each participants treatment period, up to three months.
Groups:
- Coenzyme Q and Pulmonary Hypertension: Pulmonary Hypertension subjects Nutritional Supplement Coenzyme Q-10: Nutritional Supplement
- Coenzyme Q and Healthy Controls: Healthy Control subjects Nutritional Supplement Coenzyme Q-10: Nutritional Supplement
Arm/Group | Coenzyme Q and Pulmonary Hypertension | Coenzyme Q and Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 1/10 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coenzyme Q and Pulmonary Hypertension (N=10) | Coenzyme Q and Healthy Controls (N=8)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient experienced nausea when taking Co-Q
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Length of the trial and number of subjects enrolled were both study limitations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes